CLINICAL TRIAL: NCT03537859
Title: Effect of Augmented Reality Books on Cortisol Levels in Hospitalized Pediatric Patients: a Cross-over Study.
Brief Title: Effect of Augmented Reality Books on Cortisol Levels in Hospitalized Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SIDISI 101432; 036-018 (Other: Hospital Cayetano Heredia)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Hospitalized Child
Keywords: hospitalized child; salivary cortisol; augmented reality

STUDY DESIGN:
Intervention Model Description: After enrollment, patients will be allocated in either the AR group or the NoAR group. The order of the intervention will be randomly selected before recruitment. A 48 hour wash-out will take place before the second intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality (AR) (Experimental): Books with augmented reality plus an electronic tablet.
  Interventions: Other: Augmented Reality
- Non Augmented Reality (NoAR) (Other): Conventional children book. No electronic device will be given to children.
  Interventions: Other: Non Augmented Reality

INTERVENTIONS:
Other: Augmented Reality — Augmented reality children books. The books will have special markers. The device's camera will read the marker and show 2d and 3D animations with the book's theme.
  Arms: Augmented Reality (AR)
Other: Non Augmented Reality — Augmented reality book without electronic device. Since no electronic device will be provided, the children will not be able to see any augmented reality features of the book, making it a conventional children's book.
  Arms: Non Augmented Reality (NoAR)

SUMMARY:
Hospitalization is a stressful event that might impact in a patient's recovery. Children are more susceptible to suffer acute stress as a result of a hospital stay. Stress is often quantized using cortisol levels, a substance which increases following stressful stimuli. Since stress management is important in a patient's recovery, different therapies are used and have been evaluated and proven effective to diminish cortisol levels such as play interventions and clown therapy. Nevertheless, they rely on volunteers or trained staff to perform them. Nowadays, technology such as augmented reality allow us to provide therapy without the need of volunteers. This project aims to test if augmented reality technology is effective in lowering salivary cortisol levels in hospitalized children.

DETAILED DESCRIPTION:
Background: Acute stress produced by hospitalization has a direct impact on the patient's recovery. Increased cortisol levels, the biomarker of stress, have been associated to poor health outcomes, especially on pediatric patients. Stress management in the hospital environment is essential to lower the effects of hospitalization but tend to require volunteers or other trained staff. With the advent of augmented reality technologies, providing ludic therapies to children without the need of personnel is possible. Augmented reality (AR) consists in overlapping digital information over physical objects or places creating an unique experience and the possibility of the user to interact with the technology. AR has been used in psychological and physical therapy with notable results. AR books are available in the market and are seen as a great educational tool for children. The aim of this study is to assess the effectiveness of AR books as a stress management tool in the hospital environment in a randomized cross-over study.

Sample size: Calculated taking as reference cortisol values reported previously in hospitalized children in the morning. With a 90% power and a α value of 0.05, a a significant difference of 30% of the value before the intervention is expected. For this, a sample size of 28 participants will be necessary.

Recruitment: Study participants will be recruited and enrolled in the Pediatrics Department of Cayetano Heredia Hospital. After signed consent by parents and written assent by each participant, an envelope with a random code will be opened. This code will have information of which intervention will be performed first. For AR intervention, a book and an electronic tablet will be given to the participant, for the non AR intervention (NoAR) only a book will be given. The book at the first intervention will be different than the book at the second intervention. Salivary samples will be collected before and after the intervention and a visual analogue scale (VAS) will be given to children to self-assess mood. After a 48 hour wash-out, the second intervention will take place.

Statistical analysis plan: The decrease in cortisol levels will be calculated for each participant and for each treatment. The difference in the reduction (DIF) of AR group vs. NoAR will also be calculated. A simple linear regression model will be used with DIF as dependent variable, the independent variable will be the order of intervention. The intercept will be the average decrease difference and the confidence interval will establish the statistical significance. For the secondary outcomes, the VAS will be associated with salivary cortisol.

Plan for missing data: All missing data will be reported as such.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls aged 7 - 11
* In appropriate conditions to read a book
* Hospitalization ≥ 3 days
* Capable of reading in Spanish.
* Written assent and informed consent signed by parents

Exclusion Criteria:

* Patients with adrenal diseases such as Cushing's or Addison Disease
* Patients with steroid prescription

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Change in salivary cortisol levels | Salivary samples will be obtained before and after the 1 hour intervention and kept under -20ºC until collection of samples of all participants.
  Cortisol of salivary samples will be analyzed with a commercial Enzyme Immune Assay kit (DRG , Germany).

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | VAS will be given immediately after salivary collection.
  A pictograph scale, caricatures of children with different mood going from 1 (crying) to 5 (very happy) given to children to self - assess mood.

CONTACTS AND LOCATIONS:
Overall Officials: Dulce E. Alarcón-Yaquetto, BSc, Principal Investigator — Universidad Peruana Cayetano Heredia; Cesar P Cárcamo, MD PhD, Study Director — Universidad Peruana Cayetano Heredia
Locations (1):
- Hospital Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol in spanish and english will be available. As well as the Statistical Analysis Plan and the informed consent and assent forms (in spanish)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 15, 2018
Access Criteria: Open Access
URL: https://osf.io/5q8ha/

REFERENCES:
- [Background] Bsiri-Moghaddam K, Basiri-Moghaddam M, Sadeghmoghaddam L, Ahmadi F. The concept of hospitalization of children from the view point of parents and children. Iran J Pediatr. 2011 Jun;21(2):201-8. PMID 23056788
- [Background] Mindru DE, Stanescu RS, Mioara CM, Duceac LD, Rugina A, Temneanu OR, Ungureanu M, Florescu L. STRESS IN PEDIATRIC PATIENTS--THE EFFECT OF PROLONGED HOSPITALIZATION. Rev Med Chir Soc Med Nat Iasi. 2016 Apr-Jun;120(2):417-23. PMID 27483728
- [Background] Potasz C, De Varela MJ, De Carvalho LC, Do Prado LF, Do Prado GF. Effect of play activities on hospitalized children's stress: a randomized clinical trial. Scand J Occup Ther. 2013 Jan;20(1):71-9. doi: 10.3109/11038128.2012.729087. Epub 2012 Oct 18. PMID 23078405
- [Background] Saliba FG, Adiwardana NS, Uehara EU, Silvestre RN, Leite VV, Faleiros FT, Padovani FH, De Gobbi JI. Salivary Cortisol Levels: The Importance of Clown Doctors to Reduce Stress. Pediatr Rep. 2016 Mar 31;8(1):6188. doi: 10.4081/pr.2016.6188. eCollection 2016 Mar 31. PMID 27114816
- [Background] Berryman DR. Augmented reality: a review. Med Ref Serv Q. 2012;31(2):212-8. doi: 10.1080/02763869.2012.670604. PMID 22559183
- [Background] Chicchi Giglioli IA, Pallavicini F, Pedroli E, Serino S, Riva G. Augmented Reality: A Brand New Challenge for the Assessment and Treatment of Psychological Disorders. Comput Math Methods Med. 2015;2015:862942. doi: 10.1155/2015/862942. Epub 2015 Aug 3. PMID 26339283
- [Background] McCarthy AM, Hanrahan K, Kleiber C, Zimmerman MB, Lutgendorf S, Tsalikian E. Normative salivary cortisol values and responsivity in children. Appl Nurs Res. 2009 Feb;22(1):54-62. doi: 10.1016/j.apnr.2007.04.009. PMID 19171296
- [Derived] Alarcon-Yaquetto DE, Tincopa JP, Guillen-Pinto D, Bailon N, Carcamo CP. Effect of augmented reality books in salivary cortisol levels in hospitalized pediatric patients: A randomized cross-over trial. Int J Med Inform. 2021 Apr;148:104404. doi: 10.1016/j.ijmedinf.2021.104404. Epub 2021 Feb 4. PMID 33581476